CLINICAL TRIAL: NCT05536817
Title: Prevalence of Sleep Disorder in Inflammatory Bowel Disease and Its Association With Disease Activity
Brief Title: Sleep Disorder in Inflammatory Bowel Disease and Its Association With Disease Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Julajak Limsrivilai, Associate professor, Mahidol University
Other Study IDs: SI101/2021
Record Dates: First submitted 2022-08-29; First posted 2022-09-13 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Sleep Disorder; Inflammatory Bowel Diseases
MeSH Terms: conditions — Sleep Wake Disorders; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recently, an association between active inflammatory bowel disease (IBD) and poor sleep quality has been proposed; however, the causal relationship has not yet been established. This study aimed to investigate prevalence of poor sleep quality in IBD and association with disease activity by subjective and objective measures.

Prospective observational study is conducted with expected sample size of 100 patients. Participants are classified into active and inactive disease status according to standard IBD severity assessment measures. Demographic data, disease activity, quality of life, sleep questionnaire (validated PSQI questionaire), and seven-day sleep data acquired from ambulatory wrist actigraphy were obtained. Association between sleep quality and disease activity will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed inflammatory bowel disease, followed up in Siriraj hospital, Mahidol University

Exclusion Criteria:

* Unstable medical conditions
* Known psychiatric disease
* Patients who could not withhold sedative drugs
* Pregnant patients
* Obese patients with body mass index (BMI) ≥ 35 kg/m2
* Refuse to sign a consent/ had cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over 18 years of age diagnosed with inflammatory bowel disease, either UC or CD. In addition, patients with non-IBD-related conditions that potentially impacted sleep quality will be excluded
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Subjective sleep quality | 12 months
  PSQI (Pittsburg sleep questionaire index) scores at first day then every month. PSQI contains ten questions, scoring provides sleep duration, latency, disturbance, efficiency, and quality. Total PSQI score of > 5 indicates poor sleep quality.
Objective sleep quality | 12 months
  Sleep efficiency (percentage of total sleep time compared to time-in-bed) provided by ambulatory wrist actigraphy on first seven consecutive days and at 12-month period. Score less than 85% is considered poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology division, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No